CLINICAL TRIAL: NCT07110831
Title: Influence of Fluoxetine on the Disposition Kinetics of Dolutegravir Among People Living With HIV With Major Depression in Nigeria
Brief Title: Disposition Kinetics of Dolutegravir Among People Living With HIV With Major Depression in Nigeria
Acronym: FLUDOPRESS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ibadan (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); State University of New York at Buffalo (Other); Roswell Park Cancer Institute (Other); College of Medicine University of Ibadan (Unknown); University College Hospital, Ibadan, Nigeria (Unknown); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Waheed Adeola Adedeji, Lecturer, University of Ibadan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UI/EC/22/0242; K43TW011995 (NIH)
Record Dates: First submitted 2025-05-15; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Depression; HIV
Keywords: Depression; Depressive Disorder, Major; HIV; Antidepressive Agents; Selective Serotonin Reuptake Inhibitors; Fluoxetine; Antiretroviral Therapy, Highly Active; Dolutegravir; Pharmacokinetics
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Fluoxetine; Cognitive Behavioral Therapy; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fluoxetine Arm (Experimental): Participants with a HAM-D score greater than 13 (moderate, moderately severe, and severe depression) will be recruited and allocated to the intervention group. The psychiatrist will commence the participants on fluoxetine (starting with 20mg daily). The psychiatrist will determine the dose of fluoxetine, and the dose may be adjusted during follow-up. Participants will receive Cognitive Behavioural Therapy (CBT) delivered by a Clinical psychologist in addition to fluoxetine as part of the standard routine care.
  Interventions: Drug: Fluoxetine; Behavioral: Cognitive-behavioral therapy
- Cognitive Behavioural Therapy (CBT) Arm (Active Comparator): Participants with HAM-D score between 8 and 13 (mild depression) will be recruited and allocated to the control group. They will receive only Cognitive Behavioural Therapy (CBT) as per standard routine care.
  Interventions: Behavioral: Cognitive-behavioral therapy

INTERVENTIONS:
Drug: Fluoxetine — Participants in the intervention arm will receive oral fluoxetine capsules starting with 20mg daily for 12 weeks. The dose of the fluoxetine may be adjusted during follow-up by titrating the dose against the participants' response..
  Other Names: Prozac; Fluoxetine hydrochloride; Rapiflux; Sarafem; Selfemra; Fluoxetin; Lilly-110140; N-Methyl-gamma-(4-(trifluoromethyl)phenoxy)benzenepropanamine
  Arms: Fluoxetine Arm
Behavioral: Cognitive-behavioral therapy — Participants with HAM-D score of between 8 and 13 (mild depression) will receive sessions of Cognitive Behavioural Therapy (CBT) as per standard routine care. Participants in the intervention arm will also receive sessions of CBT as per standard routine care.
  Other Names: Psychotherapy; Cognitive Behavioral Therapy; Cognitive Behavioural Therapy; Cognitive Psychotherapy; Cognitive Therapy; CBT

SUMMARY:
The goal of this clinical trial is to find out the usefulness and well-being of people when drugs for treating depression (fluoxetine) and HIV (dolutegravir) are used together. It will also learn about how safe it is to take fluoxetine and dolutegravir together by the people living with HIV (PLWH).

The main questions it aims to answer are:

* Does fluoxetine (antidepressant) make participants taking anti-HIV (dolutegravir) feel better?
* What medical problems do participants have when taking fluoxetine and dolutegravir together?
* Does what people inherit from their parents affect the effectiveness and medical problems that participants have when taking fluoxetine and dolutegravir together? Researchers will compare depression treatments, fluoxetine and psychological treatment [cognitive behavioural therapy (CBT)] together to psychological treatment (CBT) alone among adults PLWH on anti-HIV drug (dolutegravir).

Participants on anti-HIV dolutegravir having depression will:

* Take both fluoxetine (daily) and CBT together or CBT alone for 3 months
* Visit the clinic once every week in the first month, then once every 2 weeks for checkups and tests including blood tests
* Keep a diary of their symptoms and other complaints

DETAILED DESCRIPTION:
Depression is the most mental health disorder disorder among people living with HIV (PLWH) and is predictive of increased HIV-related morbidity and mortality. Treatment of depression in the setting of HIV is challenging as adding antidepressants in combination with combination antiretroviral therapy (cART) increases the pill burden and the potential for drug interactions. Studies have reported HIV medication complexity in patients comorbid with major depression to affect cART adherence. Optimal depression control among PLWH predicts and improves cART adherence and treatment outcomes.

Expert consensus is that selective serotonin-reuptake inhibitors (SSRIs) should be the first-line treatment for depression among PLWH. However, it is unclear whether SSRI therapy is effective in PLWH in low-middle-income countries (LMICs). There is an underrepresentation of LMICs in clinical studies involving PLWH and major depression despite the higher burden of PLWH and depression in LMICs than the high-income countries (HICs).

Fluoxetine is the preferred SSRI and most used for the treatment of depression in LMICs and is approved by their drug regulatory authorities. Fluoxetine is the most evaluated SSRI among PLWH with major depression but with different response rates among various ethnic groups reported. Furthermore, while fluoxetine was the most common SSRI used among the available clinical studies among PLWH, the studies did not report the clinical outcomes related to HIV care and cART.

Dolutegravir (DTG), an integrase strand transfer inhibitor, is the preferred and recommended first-line antiretroviral agent for adults and adolescents with HIV in LMICs. DTG is highly effective in suppressing HIV in both treatment-naive and experienced PLWHs, in addition to a low adverse effect profile and a high genetic barrier to developing drug resistance.

The cytochrome P450 (CYP) enzyme system metabolises fluoxetine, while the major enzyme that metabolises DTG is UGT1A1, with some contribution from CYP3A4/5. Fluoxetine and its major metabolite, norfluoxetine, may inhibit multiple enzymes involved in DTG metabolism, especially during chronic administration. A minor interaction via a membrane transporter mechanism may also be more pronounced with chronic use through the inhibition of the P-gp-mediated transport of DTG by fluoxetine. Patients on DTG report neuropsychiatric adverse events, and there is a relationship between plasma DTG trough concentration, neuropsychiatric adverse events, and UGT1A1 single nucleotide polymorphisms (SNPs). Thus, increases in DTG trough concentrations resulting from drug interaction are a potentially important concern.

Understanding potential drug interactions when fluoxetine and DGT-based cART are co-administered together will assist in optimising the dosing regimen, reducing adverse effects, and improving treatment outcomes among PLWH with major depression. To be able to recommend DTG and fluoxetine concomitant use, a prospective study involving PLWH with major depression is proposed. This study will address key knowledge gaps in drug interactions between fluoxetine and DTG among PLWH with major depression.

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 years and above
* Willing to provide informed consent.
* Confirmed HIV positive [HIV-seropositive by Enzyme Linked Immunosorbent Assay (ELISA) and Western Blot assays]
* Willingness to receive and or continue anti-HIV therapy (DTG-based cART) & adhere to follow-up schedule
* Willing and able to comply with antidepressant medication(fluoxetine) regimen and scheduled follow-up visits
* Current depressive symptoms [Subjects with depression (HAM-D-17 score ≥ 8)]
* Adequate renal function (serum creatinine < 1.5mg/dl)
* Adequate liver function [aspartate aminotransferase (AST) and alanine transaminase (ALT) ≤1.5 x Upper Limits of Normal)

Exclusion Criteria:

* Current substance use disorder
* Imminent risk of suicide- Acute suicidal ideation, gestures, or attempts
* Presence of psychotic symptoms or known diagnosis of a primary psychotic disorder
* Presence of symptoms of bipolar disorder
* Currently taking antipsychotic medication
* Pregnant or willing to get pregnant or lactation
* Current or chronic medical condition that would likely preclude adherence to protocol or completion of the trial (per investigator judgment)
* Antidepressants, mood stabilisers or other neuroleptics intake within three months
* Use of drugs other than cART, especially known enzyme inducers or inhibitors
* Abnormal ECG (e.g., prolonged QT interval)
* History of intolerance to study drug (fluoxetine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-08-14 (Estimated); Primary Completion 2027-09-30 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in the Hamilton Depression Rating Scale (HAM-D) scores from baseline to 12 weeks | Baseline to the end of treatment at 12 weeks
  The total HAM-D scores provide an indication of depression and, over time, a guide to evaluate response and recovery. The higher the HAM-D scores, the higher the severity of depression. HAM-D is graded as follows None 0-7 Mild 8-16 Moderate 17-23 Severe ≥ 24
Mean changes in the AUC of dolutegravir | Week 2 to the end of treatment at 12 weeks
  The effect of chronic administration of fluoxetine on the steady-state pharmacokinetics of dolutegravir and by intrasubject comparison in the participants. This will be assessed with mean changes in the Area under the plasma concentration-time curve (AUC) before and after the administration of fluoxetine.
Mean changes in the Cmax of doultegravir | Week 2 to the end of treatment at 12 weeks
  The effect of chronic administration of dolutegravir on the steady-state pharmacokinetics of fluoxetine by intrasubject comparison in the participants. This will be assessed with mean changes in the Maximum plasma concentration (Cmax) before and after the administration of fluoxetine.
Mean changes in the Cmin of dolutegravir | Week 2 to the end of treatment at 12 weeks
  Description: The effect of chronic administration of fluoxetine on the steady-state pharmacokinetics of dolutegravir and by intrasubject comparison in the participants. This will be assessed with mean changes in the Minimum plasma concentration(Cmin) before and after the administration of fluoxetine.
Mean changes in the AUC of fluoxetine | Week 2 to the end of treatment at 12 weeks
  The effect of chronic administration of dolutegravir on the steady-state pharmacokinetics of fluoxetine by intrasubject comparison in the participants. This will be assessed with mean changes in the Area under the plasma concentration-time curve (AUC) before and after the administration of fluoxetine.
Mean changes in the Cmax of fluoxetine | Week 2 to the end of treatment at 12 weeks
  The effect of chronic administration of dolutegravir on the steady-state pharmacokinetics of fluoxetine by intrasubject comparison in the participants. This will be assessed with mean changes in the Maximum plasma concentration (Cmax) before and after the administration of fluoxetine
Mean changes in the Cmin of fluoxetine | Week 2 to the end of treatment at 12 weeks
  The effect of chronic administration of dolutegravir on the steady-state pharmacokinetics of fluoxetine by intrasubject comparison in the participants. This will be assessed with mean changes in the Minimum plasma concentration (Cmin) before and after the administration of fluoxetine.

SECONDARY OUTCOMES:
Proportion of participants reporting grade 3 or 4 Adverse Events as Assessed by the DAIDS AE Grading Table Corrected Version 2.1 | Baseline to weeks 2, 4, 8, and 12
  The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events Corrected version 2.1 consists of parameters, or Adverse Events (AEs), with severity grading guidance that is used in DAIDS clinical trials for safety data reporting to maintain accuracy and consistency in the evaluation of AEs. The DAIDS AEs is graded as follows: Grade 1 mild event, Grade 2 moderate event, Grade 3 severe event, Grade 4 potentially life-threatening event and Grade 5 death
Proportion of participants with depression remission at week 12 | Baseline to the end of treatment at 12 weeks
  To determine the proportion of participants with depression remission at week 12 This will be measured as the proportion of subjects with HAM-D score of less than 8 (HAM-D<8)
Proportion of participants with a change of greater than or equal to (≥) 50% in the depression score from baseline to weeks 6, 8, and 12 | Baseline to weeks 6, 8 and 12
  To determine the proportion of participants with a change of greater than or equal to (≥) 50% in the HAM-D scores from baseline to weeks 6, 8 and 12
Proportion of participants that drop out (study dropouts) during the study | Baseline to weeks 2, 4, 6, 8, and 12
  To determine that proportion of participants that drop out (study dropouts) from baseline till the end of study at week 12.
Proportion of participants with viral suppression (≤ 50 copies/mL) | Baseline to the end of study at week 12
  To determine the proportion of participants with HIV viral suppression ( viral load ≤ 50 copies/mL) at the end of study at week 12
Mean increase in the CD4 count of participants | Baseline to the end of study at week 12
  To determine the mean changes in the CD4 counts of participants from baseline to the end of study at week 12
AUC of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the Area under the plasma concentration-time curve (AUC) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Cmax of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the Maximum plasma concentration (Cmax) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Cmin of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the Area Minimum plasma concentration (Cmin) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Tmax of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the time to maximum observed plasma concentration (Tmax) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Half-life (t1/2) of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the elimination half-life (t1/2) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Apparent Total Body Clearance (CL/F) of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the Apparent Total Body Clearance (CL/F) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
Apparent Volume of Distribution (Vd/F) of of fluoxetine and norfluoxetine | Weeks 2, 6,10 and 12
  To determine the Apparent Volume of Distribution (Vd/F) of fluoxetine and norfluoxetine using intensive and sparse pharmacokinetic sampling at steady state.
AUC of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Area under the plasma concentration-time curve (AUC) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Cmax of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Maximum plasma concentration (Cmax) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Cmin of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Minimum plasma concentration (Cmin) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Tmax of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Time to maximum observed plasma concentration (Tmax) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Half-Life (t1/2) of dolutegravir | Weeks 2, 6,10 and 12
  To determine the elimination Half-Life (t1/2) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Apparent Total Body Clearance (CL/F) of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Apparent Total Body Clearance (CL/F) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.
Apparent Volume of Distribution (Vd/F) of dolutegravir | Weeks 2, 6,10 and 12
  To determine the Apparent Volume of Distribution (Vd/F) of dolutegravir using intensive and sparse pharmacokinetic sampling at steady state.

CONTACTS AND LOCATIONS:
Overall Officials: Waheed A Adedeji, Principal Investigator — College of Medicine, University of Ibadan, Nigeria
Locations (1):
- University College Hospital, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data will be shared post-trial as per NIH and the University of Ibadan's policies.
Supporting Information: SAP, ICF, CSR, Analytic Code
Time Frame: After the study
Access Criteria: Researchers can access individual participant data by submitting a proposal and data sharing agreement to the principal investigator.

REFERENCES:
- [Result] Adedeji WA, Ma Q, Raji AM, Cha R, Rasaki OM, Hutson A, Taiwo BO, Charurat ME, Yusuf OB, Fehintola FA, Gureje O, Morse GD. Prevalence of depression among people living with HIV in rural hospitals in South-Western Nigeria-Association with clinico-demographic factors. AIDS Res Ther. 2023 Dec 16;20(1):89. doi: 10.1186/s12981-023-00586-0. PMID 38104102
- [Result] Borghetti A, Calcagno A, Lombardi F, Cusato J, Belmonti S, D'Avolio A, Ciccarelli N, La Monica S, Colafigli M, Delle Donne V, De Marco R, Tamburrini E, Visconti E, Di Perri G, De Luca A, Bonora S, Di Giambenedetto S. SLC22A2 variants and dolutegravir levels correlate with psychiatric symptoms in persons with HIV. J Antimicrob Chemother. 2019 Apr 1;74(4):1035-1043. doi: 10.1093/jac/dky508. PMID 30561642
- [Result] Charlier C, Broly F, Lhermitte M, Pinto E, Ansseau M, Plomteux G. Polymorphisms in the CYP 2D6 gene: association with plasma concentrations of fluoxetine and paroxetine. Ther Drug Monit. 2003 Dec;25(6):738-42. doi: 10.1097/00007691-200312000-00014. PMID 14639062
- [Result] Reese MJ, Savina PM, Generaux GT, Tracey H, Humphreys JE, Kanaoka E, Webster LO, Harmon KA, Clarke JD, Polli JW. In vitro investigations into the roles of drug transporters and metabolizing enzymes in the disposition and drug interactions of dolutegravir, a HIV integrase inhibitor. Drug Metab Dispos. 2013 Feb;41(2):353-61. doi: 10.1124/dmd.112.048918. Epub 2012 Nov 6. PMID 23132334
- [Result] Wagner GJ, Maguen S, Rabkin JG. Ethnic differences in response to fluoxetine in a controlled trial with depressed HIV-positive patients. Psychiatr Serv. 1998 Feb;49(2):239-40. doi: 10.1176/ps.49.2.239. PMID 9575014
- [Result] Yagura H, Watanabe D, Kushida H, Tomishima K, Togami H, Hirano A, Takahashi M, Hirota K, Ikuma M, Kasai D, Nishida Y, Yoshino M, Yamazaki K, Uehira T, Shirasaka T. Impact of UGT1A1 gene polymorphisms on plasma dolutegravir trough concentrations and neuropsychiatric adverse events in Japanese individuals infected with HIV-1. BMC Infect Dis. 2017 Sep 16;17(1):622. doi: 10.1186/s12879-017-2717-x. PMID 28915895
- [Result] Fettiplace A, Stainsby C, Winston A, Givens N, Puccini S, Vannappagari V, Hsu R, Fusco J, Quercia R, Aboud M, Curtis L. Psychiatric Symptoms in Patients Receiving Dolutegravir. J Acquir Immune Defic Syndr. 2017 Apr 1;74(4):423-431. doi: 10.1097/QAI.0000000000001269. PMID 27984559
- [Result] Eshun-Wilson I, Siegfried N, Akena DH, Stein DJ, Obuku EA, Joska JA. Antidepressants for depression in adults with HIV infection. Cochrane Database Syst Rev. 2018 Jan 22;1(1):CD008525. doi: 10.1002/14651858.CD008525.pub3. PMID 29355886
- [Result] Lofgren SM, Nakasujja N, Boulware DR. Systematic Review of Interventions for Depression for People Living with HIV in Africa. AIDS Behav. 2018 Jan;22(1):1-8. doi: 10.1007/s10461-017-1906-3. PMID 28900756
- [Result] Kumar V, Encinosa W. Effects of HIV Medication Complexity and Depression on Adherence to HIV Medication. Patient. 2010 Mar 1;3(1):59-69. doi: 10.2165/11531090-000000000-00000. PMID 22273276
- [Result] Egbe CO, Dakum PS, Ekong E, Kohrt BA, Minto JG, Ticao CJ. Depression, suicidality, and alcohol use disorder among people living with HIV/AIDS in Nigeria. BMC Public Health. 2017 Jun 2;17(1):542. doi: 10.1186/s12889-017-4467-5. PMID 28577548
- [Result] Obadeji A, O Ogunlesi A, O Adebowale T. Prevalence and Predictors of Depression in People living with HIV/AIDS Attending an Outpatient Clinic in Nigeria. Iran J Psychiatry Behav Sci. 2014 Spring;8(1):26-31. PMID 24995027
- [Result] Nakimuli-Mpungu E, Bass JK, Alexandre P, Mills EJ, Musisi S, Ram M, Katabira E, Nachega JB. Depression, alcohol use and adherence to antiretroviral therapy in sub-Saharan Africa: a systematic review. AIDS Behav. 2012 Nov;16(8):2101-18. doi: 10.1007/s10461-011-0087-8. PMID 22116638
- [Result] Brown GR, Rundell JR, McManis SE, Kendall SN, Zachary R, Temoshok L. Prevalence of psychiatric disorders in early stages of HIV infection. Psychosom Med. 1992 Sep-Oct;54(5):588-601. doi: 10.1097/00006842-199209000-00006. PMID 1438661
- [Result] Arseniou S, Arvaniti A, Samakouri M. HIV infection and depression. Psychiatry Clin Neurosci. 2014 Feb;68(2):96-109. doi: 10.1111/pcn.12097. Epub 2013 Oct 30. PMID 24552630
- [Result] Satz P, Myers HF, Maj M, Fawzy F, Forney DL, Bing EG, Richardson MA, Janssen R. Depression, substance use, and sexual orientation as cofactors in HIV-1 infected men: cross-cultural comparisons. NIDA Res Monogr. 1997;172:130-55. No abstract available. PMID 9154269